CLINICAL TRIAL: NCT00072579
Title: Phase II Study of GM-CSF in Patients With Chronic Phase Chronic Myeloid Leukemia (CP-CML) Who Are Not in Complete Cytogenetic Remission After Initial Therapy
Brief Title: Sargramostim in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia Who Are Not in Complete Cytogenetic Remission Following Initial Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU-23102; CDR0000340983 (Registry Identifier: PDQ (Physician Data Query)); BRLX-02153; NCI-7350
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — sargramostim

INTERVENTIONS:
Biological: sargramostim

SUMMARY:
RATIONALE: Colony-stimulating factors, such as sargramostim, may increase the number of immune cells found in bone marrow or peripheral blood and may bring about complete remission in patients who have chronic phase chronic myelogenous leukemia.

PURPOSE: This phase II trial is studying sargramostim to see how well it works in treating patients with chronic phase chronic myelogenous leukemia that is not in complete cytogenetic remission after initial treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and safety of sargramostim (GM-CSF) by cytogenetic examination of the bone marrow in patients with chronic phase chronic myelogenous leukemia who are not in complete cytogenetic remission after initial therapy.

OUTLINE: Patients receive sargramostim (GM-CSF) subcutaneously daily for 3 months in the absence of disease progression or unacceptable toxicity. Patients achieving no response receive GM-CSF for an additional 3 months. Patients failing to achieve a partial response or better after the second course of GM-CSF are removed from the study. Patients achieving a partial response after the first or second course of GM-CSF continue to receive GM-CSF for an additional 9 months. Patients are then re-evaluated. Patients achieving a complete cytologic response at 9 months then receive GM-CSF 3 times weekly in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 weeks.

PROJECTED ACCRUAL: A total of 9-24 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed chronic phase chronic myelogenous leukemia (CML)

  * Presence of t(9;22)(q34;q11) with at least 20 cells examined in metaphase by cytogenetic examination of the bone marrow
* Complete hematologic remission during prior therapy* as seen on 2 separate blood count analyses, defined by the following:

  * WBC no greater than 10,000/mm^3 AND platelet count no greater than 450,000/mm^3
  * Disappearance of all signs and symptoms of disease, including palpable splenomegaly
  * Normal differential counts (i.e., absence of blasts, promyelocytes, myelocytes, and metamyelocytes) NOTE: *Continuation of therapy that led to complete hematologic remission is required during study participation
* Persistent cytogenetic disease despite 12 months of prior imatinib mesylate therapy, which may have included a trial dose-escalation OR intolerant of imatinib mesylate at a dose greater than 400 mg/day
* Not in complete cytogenetic remission within 30 days of study entry

  * Persistent Philadelphia chromosome by bone marrow exam

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled active infective
* No serious medical or psychiatric illness that would prevent giving informed consent or limit survival to less than 6 months
* No other malignancy not in remission except curatively treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior sargramostim (GM-CSF) allowed
* Prior interferon alfa for CML allowed
* No prior stem cell transplantation
* Concurrent interferon alfa* for CML allowed NOTE: *No dose increase during study participation

Chemotherapy

* At least 4 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 4 weeks since prior surgery

Other

* Prior imatinib mesylate for CML allowed
* No other concurrent medication for CML
* Concurrent imatinib mesylate* for CML allowed NOTE: *No dose increase during study participation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2006-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cytogenetic response (complete and partial)

SECONDARY OUTCOMES:
Toxicity as assessed by the Expanded Common Toxicity Criteria v2.0
Time to progression
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Molnar, MD, Study Chair — Wake Forest University Health Sciences; Bayard L. Powell, MD — Wake Forest University Health Sciences
Locations (15):
- United States (15):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - CCOP - Central Illinois, Decatur, Illinois
  - Kentuckiana Cancer Institute, PLLC, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Alamance Cancer Center, Burlington, North Carolina
  - Hugh Chatham Memorial Hospital, Elkin, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina